CLINICAL TRIAL: NCT05388461
Title: Acute Efficacy and 6 Months Follow up After Electroconvulsive Therapy for Severe or Treatment Resistant Depression - Predictors of Response, Side Effects, and Relapse
Brief Title: Acute Efficacy and 6 Months Follow up After Electroconvulsive Therapy
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018/2541
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Electroconvulsive Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: electroconvulsive therapy — electroconvulsive therapy

SUMMARY:
The overall aim of the current project is to assess the acute and long term outcome of ECT (both patient and clinician rated) in a non-selected patient cohort from ordinary clinical activity, and to seek out factors predicting response and remission, side effects and relapse.

DETAILED DESCRIPTION:
Patients reffered to electroconvulsive ECT are (after written consent) enroled in a research registry. Based on (clinician and patient rated) measures of depressive symptoms and overall cognitive function, the short and long-term (6 months) efficacy of ECT will be described, and factors predicting response and relapse identified.

The duration of possible cognitive impairment and factors predicting cognitive outcome will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with ECT for major depression (F31.3-5, F32, F33) at Haukeland University Hospital or Stavanger University Hospital after 2013,
* written consent to enrolment into the Regional Register for neurostimulation.

Exclusion Criteria:

* ECT performed on other indications than major depression.
* No consent to the register.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: population based cohort from ordinary clinical activity
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-03-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of Montgomery and Åsberg Depression Rating Scale (MADRS) score from pretreatment at posttreatment; MADRS range 0 - 60, with higher scores indicating more severe depression) | up to 8 weeks
  depressive symptoms
Change of Mini Mental State Examination (MMSE-NR) score from pretreatment at posttreatment; MMS-E range 0-30 with lower scores indicating more severe cognitive impairment | up to 8 weeks
  overall cognitive function
Change of Beck depression inventory (BDI) score from pretreatment at posttreatment; BDI range 0-63, with higher scores indicating more severe depression | up to 8 weeks
  depressive symptoms, patient rated
Change of Everyday Memory Questionnaire (EMQ) score from pretreatment at posttreatment with higher scores indicating more severe impairment | up to 8 weeks
  overall subjective cognitive function, patient rated

SECONDARY OUTCOMES:
Change of Patient rated improvement (PGI) score from pretreatment at posttreatment | up to 8 weeks
  Likert scale
Change of Clinical Global Impression (CGI) score from pretreatment at posttreatment | up to 8 weeks
  Likert scale
Change of Subjective cognitive function score from pretreatment at posttreatment | up to 8 weeks
  Likert scale
Change of Montgomery and Åsberg Depression Rating Scale (MADRS) score from pretreatment at follow up, MADRS range 0 - 60, with higher scores indicating more severe depression) | 6 months
  depressive symptoms
Change of Mini Mental State Examination (MMSE-NR) score from pretreatment at follow up, MMS-E range 0-30 with lower scores indicating more severe cognitive impairment | 6 months
  overall cognitive function
Change of Beck depression inventory (BDI) score from pretreatment at follow up, BDI range 0-63, with higher scores indicating more severe depression | 6 months
  depressive symptoms, patient rated
Change of Everyday Memory Questionnaire (EMQ) score from pretreatment at follow up | 6 months
  overall subjective cognitive function, patient rated
Change of Patient rated improvement (PGI) score from pretreatment at follow up | 6 months
  Likert scale
Change of Clinical Global Impression scale (CGI) from pretreatment at follow up | 6 months
  Likert scale

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger

IPD SHARING:
Plan to Share IPD: Undecided
after approval from data protection manager IPD will be shared on reasonable request